CLINICAL TRIAL: NCT05928923
Title: The Screening and the Treatment of ECG Holter and Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202003021RIPB
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-04

CONDITIONS: The Screening and the Treatment of ECG Holter and Sleep Apnea
Keywords: sleep healthcare; actigraph devices; questionnaires; ECG Holter
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cpap (Experimental): usage cpap 3 months
  Interventions: Device: CPAP
- Usual care (No Intervention): Usual care 3smonths

INTERVENTIONS:
Device: CPAP — CPAP usage 3 months
  Arms: cpap

SUMMARY:
Sleep quality affect working and learning performance; poor quality of sleep is one of the common problems of modern people. Traditionally, polysomnography is a recognized standard for sleep quality assessment. Subjects are put adhesive electrodes, chest and abdomen band, oximetery, and oronasal cannula and stay in certified sleep laboratory for monitoring. These sensors setup are cumbersome and be likely to induce discomfort. An alternative to assess the quality of sleep is actigraphy, which allows users to wear for more than two weeks. In recent years, many of the devices, which often measure physiological signals, are prevailing to make long-term sleep monitoring feasible, but its accuracy and effectiveness still need to be verified.

Obstructive sleep apnea (OSA) is a common disorder characterized by intermittent hypoxia and sleep fragmentation. OSA is associated with cardiovascular morbidity and mortality, metabolic dysregulation, and neurocognitive dysfunction, which results in the negative impact on prognosis. PSG is the gold standard for OSA diagnosis which is expensive and less accessible. Therefore, modality other than PSG is necessary to speed up diagnosis and treatment. Center of Sleep Disorder in National Taiwan University Hospital has been operated since June 2006. Up to Dec.2015, totally 8,819 patients have been referred for sleep studies (NTUH cohort) where 1,435 patients are under long-term CPAP and 396 patients are under MAD. Using data from 4,618 patients in NTUH cohort, we have already established an OSA prediction mode (apnea-hypopnea index, AHI≥5/hr) with accuracy 82.37% (sensitivity 87.03%, positive predictive value 91%). Regarding the molecular mechanism, our previous study showed that by plasma metabolomics profiling, we could identify candidate metabolites associated with OSA severity. The 11 candidate metabolites were identified by comparing profiling in 100 patients with AHI <15/hr and with AHI≥ 15/hr, respectively. Six identified metabolites were selected to establish an AHI prediction model which gave sensitivity 66%, specificity 72%, and AUROC 0.736. Furthermore, 15 plasma metabolites associated with excessive daytime sleepiness (EDS) or polysomnographic parameters were identified. Among those metabolites, L-Kynurenine and g-Glutamylleucine were metabolites associated with EDS which generated the AUROC to EDS prediction as 63% in study group and 76.7% in validation group. The "LARGAN"ECG Holter for diagnosis of sleep disorder has been set up by LARGAN-health. It aims on population with simple diagnosis of sleep disorder. Combining the "LARGAN"ECG Holter provides the diagnosis and solution of sleep disorder, sleep tracking, and education. This devices is almost set and needs the input from general population to validate the accuracy.

The trial, which includes questionnaires, Actigraph devices, 24-hr BP and "LARGAN"ECG Holter for long-term home sleep monitoring, is proposed to allow users to detect potential subjects who have sleep disorders by using the ECG Holter. The aims of the present project include: (1) All 190 voluntary. Recruit 30 voluntary participants from patients with mild OSA (AHI≥5-15/hr), 160 for each voluntary participants from patients with moderate OSA (AHI≥15-30/hr) and severe OSA (AHI≥30/hr) to validate agreement of sleep efficiency via this trial, Actigraph devices and ECG Holter for 9 days, and 24 hour blood pressure for one day. (2) All participants will take an overnight PSG test, blood sampling, basal metabolism measurement, Actigraph devices, ECG Holter, body composition and E-Prime at the sleep center to validate the performance of this system on diagnosis of OSA in low risk population. (3) Analyze the of PSG parameters in both low and high risk population (to build up the out of center devices for OSA home testing). (4) Integrate the clinical parameters and plasma metabolic profile, before and after treatment, to identify factors associated with OSA related sequels and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. age:≧20 year-old
2. Mild Obstructive Sleep Apnea (AHI≥5-15/hr)(30 patients)
3. Moderate Obstructive Sleep Apnea (AHI≥15-30/hr) (80 patients)
4. Severe Obstructive Sleep Apnea (AHI≥30/hr)(80 patients)

Exclusion Criteria:

1. skin allergy
2. wrist tattoos
3. BMI≧40 kg/m2
4. Neurological Disorders(Infection, Stroke, ALS, Myopathy, Brain tumor and Encephalitis)
5. Internal Diseases(cardiovascular disease or coronary artery disease was poorly controlled
6. chronic heart failure(including NYHA class 3 or more than NYHA class 3)
7. COPD(FEV1/FVC<70)
8. Hyperthyroidism or Hypothyroidism
9. Primary Aldosteronism
10. Chronic Kidney Disease(eGFR<30)
11. Acromegaly and Parkinson's disease)
12. Psychosis(Schizophrenia, bipolar disorder and depression)
13. Autoimmune disease(System Lupus Erythematosus, Rheumatoid arthritis, Sarcoidosis, Crohn's disease and Ulcerative Colitis)
14. Cancer(in last 5 years)
15. Have been diagnosed with obstructive sleep apnea
16. other sleep disorder(Narcolepsy, insomnia and RBD)
17. Use anti-inflammatory drugs(in last 2 weeks)
18. Illiterate
19. shift worker
20. has been Spinal Surgery and move difficult
21. professional driver has severe drowsiness

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Questionnaires from OSA population | 36 months
  Primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Center of sleep disorders, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No